CLINICAL TRIAL: NCT04586270
Title: A Phase 1 Study of TAS0612 in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of TAS0612 in Participants With Advanced or Metastatic Solid Tumor Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Taiho Oncology as the sponsor of study TAS0612-101, has made a strategic decision to terminate the TAS0612-101 study, taking into consideration the safety profile of TAS0612 and the absence of encouraging anti-tumor activity.
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAS0612-101; 2020-002304-39 (EudraCT Number)
Record Dates: First submitted 2020-09-23; First posted 2020-10-14 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Advanced or Metastatic Solid Tumors
Keywords: Solid Tumors; AKT inhibitor; RSK inhibitor; S6K inhibitor; kinase inhibitor; phase I; Prostate cancer; PTEN loss; PTEN mutation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TAS0612 Escalation (Experimental): TAS0612 administered orally
  Interventions: Drug: TAS0612
- TAS0612 Expansion (Experimental): TAS0612 administered orally
  Interventions: Drug: TAS0612

INTERVENTIONS:
Drug: TAS0612 — oral tablets

SUMMARY:
The purpose of this study is to see if TAS0612 is safe in participants with advanced or metastatic solid tumor cancer.

ELIGIBILITY:
Inclusion Criteria:

Dose Escalation:

Have histologically confirmed, locally advanced, and unresectable cancer, or metastatic cancer and have progressed on or were intolerant to standard treatments or refused standard of care (SOC).

Dose Expansion:

Have documented histologically or cytologically confirmed adenocarcinoma of the prostate with documented PTEN loss or loss of function mutation, who have metastatic castration-resistant disease and have:

* Disease progression per the Prostate Cancer Clinical Trials Working Group 3 (PCWG3)/modified RECIST 1.1 after the most recent regimen.
* Received androgen receptor directed therapy previously with or without chemotherapy consisting of no more than 2 prior taxane-based regimens.
* Been receiving androgen deprivation therapy with serum testosterone <50 ng/dL (<2.0 nM). Note: previously documented PTEN loss or loss of function mutation from archived tissue sample testing or cfDNA sample testing is acceptable if done in a CLIA certified lab or a locally certified lab.

Have an ECOG score of 0 or 1 Dose Escalation (Part 1): Have no measurable or measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

Dose Expansion (Part 2): Have measurable or no measurable disease per PCWG3/modified RECIST 1.1

• No more than 30 patients with no measurable disease will be enrolled in Dose Expansion (Part 2).

Exclusion Criteria:

* Participating in medical research not compatible with this study
* Have not discontinued or recovered from previous treatments for cancer
* Have a significant cardiac condition
* Have untreated brain metastases
* Have a primary brain tumor
* Have a serious concomitant disorder
* Unable to swallow or digest pills
* Poorly controlled diabetes
* Concomitant medications or substances that are strong inhibitors/inducers of CYP3A.Study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-11-14 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLTs) | Baseline through Cycle 1 (28-day cycle)
  Number of participants with DLTs during cycle 1
rPFS rate | Baseline through measured progressive disease (estimated up to 12 months)
  Percentage of participants with partial response (PR) or complete response (CR) at 6 months Prostate Cancer Working Group 3 (PCWG3)/ modified defined by the Response Evaluation Criteria in Solid Tumors (mRECIST) v1.1.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) per PCWG3/mRECIST1.1 | Baseline through progressive disease or date of death for any causes, whichever comes first, assessed up to 12 months.
  DCR: Percentage of participants who exhibit stable disease (SD), PR or CR.
Duration of Response (DOR) per PCWG3/mRECIST1.1 | Baseline through progressive disease or date of death for any causes, whichever comes first, assessed up to 12 months.
  DOR: Date of PR or CR to date of objective progression or death due to any cause.
Radiographic Progression Free Survival (rPFS) per PCWG3/mRECIST1.1 | Baseline through progressive disease or date of death for any causes, whichever comes first, assessed up to 6 months.
  Proportion of patients experiencing a radiographic progression by PCWG3/mRECIST1.1 criteria
Overall Response Rate (ORR) per PCWG3/mRECIST1.1 | Baseline through progressive disease or date of death for any causes, whichever comes first, assessed up to 12 months.
  Proportion of patients experiencing a best overall response of Complete Response (CR) or Partial response (PR)
Prostatic Specific Antigen (PSA) Response | Baseline to PSA progression, up to 12 months
  Proportion of patients with ≥50% reduction in PSA from baseline to lowest post-baseline result.
Pharmacokinetics (PK) parameters including but not limited to: Cmax | Cycle 1 Day 1 through Cycle 1 Day 15 (28-day cycle) Cycle 2 Day 1 and Cycle 3 Day 1
  time of TAS0612 it takes to reach Cmax.
Pharmacokinetics (PK) parameters including but not limited to: Tmax | Cycle 1 Day 1 through Cycle 1 Day 15 (28-day cycle) Cycle 2 Day 1 and Cycle 3 Day 1
  time of TAS0612 it takes to reach Cmax,
Pharmacokinetics (PK) parameters including but not limited to: AUC. | Cycle 1 Day 1 through Cycle 1 Day 15 (28-day cycle) Cycle 2 Day 1 and Cycle 3 Day 1
  Area under the plasma concentration curve of TAS0612.
Pharmacokinetics (PK) parameters including but not limited to: T1/2. | Cycle 1 Day 1 through Cycle 1 Day 15 (28-day cycle) Cycle 2 Day 1 and Cycle 3 Day 1
  time it takes for plasma concentration to fall by half its original value (t1/2) of TAS0612
Safety and Tolerability | From screening to 30 days after last dose
  All adverse events (AEs) per CTCAE v5.0.
Pharmacodynamic: biochemical effects of TAS0612: Total proteins | Cycle 1 Day 1 through Cycle 1 Day 15 (28-day cycle)
  Total proteins will be measured in blood samples collected at different time points.
Pharmacodynamic: biochemical effects of TAS0612: phospho-proteins | Cycle 1 Day 1 through Cycle 1 Day 15 (28-day cycle)
  Phospho-proteins will be measured in blood samples collected at different time points. The levels/changes (dose- and concentration-dependent) of phospho-proteins will be assessed and reported for biochemical effects of TAS0612.
Pharmacodynamic: molecular effects in tumor tissue of TAS0612 | Baseline through Day 1 Cycle 2 (28-day cycle) through study completion, an average of 1 year
  Selected phospho-proteins will be analyzed in tumor tissue at baseline and on-treatment in dose escalation. The levels/changes of the phospho-proteins will be assessed and reported for target modulation.

OTHER OUTCOMES:
Pharmacokinetics (PK): Metabolites in plasma | Cycle 1 Day 1 (each cycle is 28 days).
  Structure elucidation of TAS0612 metabolites in human plasma.
Time-matched plasma exposures of TAS0612 and changes from baseline in QTcF using central ECG measurements | Baseline through progressive disease or date of death for any causes, whichever comes first, assessed up to 12 months
  To explore the correlation between the incidence of exposures of TAS0612 in plasma and QT prolongation
Exploratory correlation of tissue and/or blood markers with tumor efficacy endpoints and/or tumor resistance to TAS0612 | Baseline through progressive disease or date of death for any causes, whichever comes first, assessed up to 12 months.
  To investigate potential predictive biomarkers for TAS0612.
Exposure of TAS0612 and selected efficacy and safety measures. | Baseline through progressive disease or date of death for any causes, whichever comes first, assessed up to 12 months.
  To explore the correlation between PK and antitumor activity or toxicity

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - Tennessee Oncology, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- France (2):
  - Institut Paoli Calmette, Marseille, Bouches Du Rhone
  - Centre de Lutte Contre le Cancer Gustave Roussy, Villejuif, Val De Marne

IPD SHARING:
Plan to Share IPD: No